CLINICAL TRIAL: NCT02295189
Title: Ketorolac Versus Triamcinolone Intra-articular Knee Injections for the Treatment of Osteoarthritis. A Prospective, Double-Blinded Randomized Trial
Brief Title: Ketorolac Versus Triamcinolone Knee Injections for Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: San Antonio Military Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Jaime L. Bellamy, DO, Orthopaedic Resident Physician, San Antonio Military Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SanAntonioMMC
Record Dates: First submitted 2014-11-12; First posted 2014-11-20 (Estimated); Last update posted 2014-11-20 (Estimated); Status verified 2014-11

CONDITIONS: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Ketorolac Tromethamine; Triamcinolone Acetonide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Visual analogue scale (Active Comparator): visual analogue scale versus triamcinolone acetonide visual analogue scale versus ketorolac tromethamine
  Interventions: Drug: Ketorolac Tromethamine; Drug: Triamcinolone Acetonide
- Treatment (Active Comparator): visual analogue scale versus triamcinolone acetonide visual analogue scale versus ketorolac tromethamine
  Interventions: Drug: Ketorolac Tromethamine; Drug: Triamcinolone Acetonide

INTERVENTIONS:
Drug: Ketorolac Tromethamine — anti-inflammatory injection
  Other Names: Toradol
Drug: Triamcinolone Acetonide — corticosteroid injection
  Other Names: Kenalog

SUMMARY:
Osteoarthritis is a disabling disease of the joint spaces and has a high impact on society due to the amount of people who are affected by the disease. Nonoperative management is a mainstay of therapy in most patients. Ketorolac tromethamine and triamcinolone acetonide intra-articular knee injections will be compared in a prospective, double-blinded, randomized trial in subjects with knee osteoarthritis. Subjects will be enrolled from the Orthopaedics Clinic based on inclusion and exclusion criteria. Intra-articular knee injection of ketorolac tromethamine or triamcinolone acetonide will be performed under ultrasound guidance. Multiple outcome measures will be performed throughout the six month period of follow-up. The investigators predict ketorolac tromethamine will have a longer duration of pain relief when compared to triamcinolone acetonide. The investigators predict there will be no differences between the two intra-articular knee injections in terms of function using validated scoring instruments.

DETAILED DESCRIPTION:
Subject Population: Adult patients, age 18-90 years old who satisfy the inclusion criteria and do not meet the exclusion criteria will be enrolled from the Orthopaedics Clinic at San Antonio Military Medical Center (SAMMC). The enrollment period for this study is two years, patients will be recruited up to 44 enrollees to allow 36 completers. Patients will be stratified based on gender and age (< 65 or >= 65 years old). Demographics obtained will be age, gender, height, weight, laterality and body-mass index (BMI).

Randomization: This will be a predetermined computerized randomization schedule to identify treatment, ketorolac tromethamine versus triamcinolone acetonide. A patient key on paper listing the patient name, last four digits of sponsor's social security number, study number (randomly assigned), and treatment will be kept with the nurse/technician in the Orthopaedics Clinic, locked in a cabinet. Patients will be stratified by gender and age (< 65 or >= 65 years old). Subjects will continue to be enrolled until there are at least 10 of each gender in each group, treated with either ketorolac tromethamine or triamcinolone acetonide. In the event the subject has bilateral knee pain, both knees will be injected with the same treatment medication and the knee will be randomized as to which one will be included in the data analysis.

A pharmacist will prepare the treatment injection in the Orthopaedics Clinic. Injections will be done with a 2-inch, 21-gauge needle placed on a 10cc syringe with an opaque covering to conceal its contents to blind the patient and associate investigator to treatment. Injections will contain either 2cc of ketorolac tromethamine (Toradol, 15mg/cc) in 8cc of bupivacaine hydrochloride (0.5%) without epinephrine or 2cc of triamcinolone acetonide (Kenalog-40, 40mg/cc) in 8cc of bupivacaine hydrochloride (0.5%) without epinephrine. The subject and the treatment injection will be taken to the Interdisciplinary Pain Management Center, for injection under ultrasound guidance. The subject's selected knee, or bilateral knees, at the superolateral site, will be sterilely prepped in standard fashion with betadine and allowed to dry, prior to injection. The treatment will be injected by the associate investigator, in the Interdisciplinary Pain Management Center, who is trained in Physical Medicine and Rehabilitation and certified to perform ultrasound examinations. The associate investigator will be blinded to treatment and outcomes.

A patient key listing the patient name, last four digits of sponsor's social security number, age, gender, patient number (randomly assigned) and treatment received will be kept with the nurse/technician in the Orthopaedics Clinic in a research folder, locked in a cabinet.

Radiographs will be obtained at baseline and at 6 months follow-up. Osteoarthritis will be classified according to Kellgren-Lawrence (K-L) radiographic criteria by associate investigator who is fellowship trained in Total Joints. K-L grading will be entered on the Case Report Form (CRF) prior to outcome data entry. The associate investigator will be blinded to treatment. Outcome data collection will be performed by a study nurse/technician in the Orthopaedics Clinic, with the exception of part of the Knee Society Score (KSS), which will be performed by an associate investigator. The nurse/technician will record demographic data, including height, weight, BMI, gender, laterality and age, at the baseline clinic visit and at the 6 month follow-up. The use of nonsteroidal anti-inflammatory drug (NSAID) and analgesic drugs and adverse events during the study period will be recorded at each visit. Patients will keep a diary of NSAID and analgesic use during the study. Patients will follow-up at 2 weeks, 6 weeks, 3 months and 6 months. A visual analogue scale (VAS), KSS, Western Ontario and McMasters Universities (WOMAC) index, Short Form 36 (SF-36), University California Los Angeles (UCLA) Activity Score and Lysholm Knee Score (LKS) will be obtained at the baseline clinic visit and each follow-up. All data obtained from the study will be recorded on the CRF. All data collected will be kept with the nurse/technician in the Orthopaedics Clinic in a research folder, locked in a cabinet.

Data from the CRF will be entered into an electronic database on Excel by the principle investigator on a password protected computer. The database will be made available to the associate investigators electronically. Data analysis will be performed by the principle investigator which will also be performed on a password protected computer. All investigators will remain blinded to the treatment received, until all data analysis is performed. There will be no patient identifiers in the data provided to the investigators, only the patient number. The patient number is a number randomly assigned to the patient and is only identifiable in the patient key, which will be kept separate as above.

A sample size of 16 per group achieve 80% power to detect a difference of 1.6 (16mm) VAS comparing ketorolac tromethamine to triamcinolone acetonide intra-articular injections with estimated standard deviations of 1.56 and with a significance level (alpha) of 0.05. There is an expected drop-out rate of 20%, which implies a sample size of 20 subjects per group. Data analysis will be performed by the principle investigator and associate investigator who will be blinded to treatment until data analysis is complete.

ELIGIBILITY:
Inclusion Criteria:

* Subject must be at least 18 years of age and no older than 90 years of age; of either gender
* Radiographic evidence of symptomatic osteoarthritis in one or bilateral knees. Osteoarthritis will be defined as pain with weight-bearing at the tibiofemoral and/or patellofemoral articulation together with radiographic findings as described below.

At the painful articulation, radiographic evidence of Kellgren-Lawrence

* Grade 2: definite osteophytes and possible narrowing of joint cartilage associated with sclerosis of subchondral bone or,
* Grade 3: moderate multiple osteophytes, definite narrowing of the joint space, small pseudocystic areas with sclerotic walls in the subchondral bone, possible deformity of bone ends or,
* Grade 4: large osteophytes, marked narrowing of joint space, severe sclerosis and altered shape of the bone ends.

Subject agrees to participate in follow-up evaluations and complete outcome score sheets (post-injection, 2 weeks, 6 weeks, 3 months and 6 months).

Exclusion Criteria:

* Any inflammatory or neuropathic arthropathy
* Insufficiency of the collateral ligaments or cruciate ligaments
* Current infection
* Recent injection (<3 months)
* Pregnant/lactating (β-human chorionic gonadotropin pregnancy test will be completed prior to injection)
* Allergy or hypersensitivity to the study medications
* Currently taking any anti-coagulation medications
* Subject is unable to make his/her own decision regarding the informed consent
* Subject is unable to read/understand English

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2013-01; Primary Completion 2014-05 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Change in Visual analogue scale (VAS) | Baseline, 2 weeks, 6 weeks, 3 months, 6 months

SECONDARY OUTCOMES:
Change in Western Ontario and McMaster Universities Index (WOMAC) | Baseline, 2 weeks, 6 weeks, 3 months, 6 months
Change in Knee Society Score (KSS) | Baseline, 2 weeks, 6 weeks, 3 months, 6 months
Change in Tegner-Lysholm Knee Score (TLK) | Baseline, 2 weeks, 6 weeks, 3 months, 6 months
Change in Short Form (SF-36) | Baseline, 2 weeks, 6 weeks, 3 months, 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Siraj Sayeed, MD, Principal Investigator — San Antonio Military Medical Center